CLINICAL TRIAL: NCT00432783
Title: A Comparison of Adherence Rates to Ritonavir (Soft-gel Capsules) and Its Accompanying Protease Inhibitor (PI) in Patients Receiving Ritonavir Boosted PI Regimens
Brief Title: A Comparison of Adherence Rates to Ritonavir and Its Accompanying Protease Inhibitor
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Jonathan Shuter, Prof. Dept Medicine, Montefiore Medical Center
Other Study IDs: 06-01-023E
Record Dates: First submitted 2007-02-06; First posted 2007-02-08 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: HIV Infections
Keywords: HIV, antiretroviral therapy, adherence, ritonavir
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Pharmacologic boosting of protease inhibitors with ritonavir has become standard practice in antiretroviral therapy. Patients are instructed to take ritonavir at the same time as its accompanying protease inhibitor. However, ritonavir is unpopular with many patients because of its large size and because of the recommended need for refrigeration. This study will test the hypothesis that adherence to ritonavir is inferior to adherence to its accompanying protease inhibitor in patients receiving such therapy.

DETAILED DESCRIPTION:
The study staff will employ MEMS caps to prospectively measure adherence to ritonavir and its accompanying protease inhibitor over 24 weeks of follow-up. Paired sample t-tests will be employed to compare adherence to the two agents, and secondary analyses will be conducted to evaluate the chronologic concordance of ritonavir and accompanying protease inhibitor dosing.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection, age>18 years, receiving therapy with ritonavir-boosted atazanavir or fosamprenavir, willingness to use MEMS caps, willingness to provide informed consent

Exclusion Criteria:

* Treatment with any medication that is contraindicated in combination with ritonavir or its accompanying protease inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from the Montefiore Medical Center Infectious Diseases Clinic who meet eligibility criteria described below.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2006-06 (Actual); Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Shuter, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Shuter J, Sarlo JA, Rode RA, Zingman BS. Occurrence of selective ritonavir nonadherence and dose-staggering in recipients of boosted HIV-1 protease inhibitor therapy. HIV Clin Trials. 2009 May-Jun;10(3):135-42. doi: 10.1310/hct1003-135. PMID 19632952